CLINICAL TRIAL: NCT03523507
Title: A Randomized, Sham-controlled, Double-blinded Study of Bilateral Prefrontal Individual Connectome-targeted Repetitive Transcranial Magnetic Stimulation to Treat the Symptoms of Depression Associated With Concussive Traumatic Brain Injury.
Brief Title: fMRI-neuronavigated rTMS Treatment for Symptoms of Depression Associated With Concussive TBI in the Military Population
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Study terminated due to COVID-19 restrictions
Sponsor: Henry M. Jackson Foundation for the Advancement of Military Medicine (Other)
Collaborators: Center for Neuroscience and Regenerative Medicine (CNRM) (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 898115
Record Dates: First submitted 2017-12-20; First posted 2018-05-14 (Actual); Last update posted 2020-11-03 (Actual); Status verified 2019-07

CONDITIONS: Traumatic Brain Injury; Concussion, Mild; Depressive Symptoms
Keywords: Repetitive Transcranial Magnetic Stimulation; Military
MeSH Terms: conditions — Brain Injuries, Traumatic; Brain Concussion; Depression

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Active: rTMS (Experimental): Participants will receive 20 bilateral treatment sessions provided over approximately a 5-week period. Daily sessions entail approximately 60 minutes of time.
  Interventions: Device: Active: rTMS
- Sham: rTMS (Sham Comparator): Sham: Repetitive Transcranial Magnetic Stimulation; Participants will receive sham treatment designed to have similar sound and tactile sensation, without producing active stimulation.
  Interventions: Device: Sham: rTMS

INTERVENTIONS:
Device: Active: rTMS — Daily sessions will consist of 3000 left-sided excitatory pulses at 10 Hz (with 4-second trains and 26-second inter-train interval) followed by 1000 right-sided inhibitory pulses at 1 Hz (in a single train). The DLPFC treatment target will be determined using individualized resting-state network mapping.
  Arms: Active: rTMS
Device: Sham: rTMS — Daily sessions will consist of the same total number of sham pulses, designed to have similar sound and tactile sensation, without producing active stimulation.
  Arms: Sham: rTMS

SUMMARY:
This study aims to investigate the efficacy and tolerability of fMRI-targeted repetitive transcranial magnetic stimulation (rTMS) in the treatment of depressive symptoms in service members with a history of concussive traumatic brain injury (TBI).

Up to ninety participants will be randomized to active or sham treatment. Participants randomized into the active group will receive 20 sessions of left-sided dorsolateral prefrontal cortex (DLFPC) high-frequency rTMS, followed by right-sided DLFPC low-frequency rTMS. The DLPFC treatment area will be identified by using individual subject-level resting state network estimation (Hacker et al., 2013). Participants randomized into the sham treatment group will receive 20 sham treatments designed to have similar sound and tactile sensation, without producing active treatment. Participants will also be asked to complete regular follow-up evaluations for up to a total of six follow-up sessions. Those who do not respond to the treatment will have the option to receive active treatment through this study regardless of group assignment to active or sham.

DETAILED DESCRIPTION:
This study aims to investigate the efficacy and tolerability of individual connectome-targeted repetitive transcranial magnetic stimulation (ICT-rTMS) treatment to enhance the rehabilitation of service members with symptoms of depression and history of concussive traumatic brain injury (TBI).

This will be a multi-site, double-blinded, sham-controlled, prospective, randomized interventional trial. Up to ninety participants will be block randomized to active (ICT-rTMS) or sham treatment. Participants will receive 20 sessions of ICT-rTMS over approximately 5 weeks.

Resting-state functional magnetic resonance imaging (rsfMRI) and structural MRI will be obtained at baseline to allow for the calculation of connectome-targeted treatment coordinates and ensure the absence of structural abnormalities. The rsfMRI scan at baseline will also be used to establish the baseline for the secondary imaging outcome measures.

Treatment sessions will consist of high-frequency left dorsolateral prefrontal cortex (DLPFC) stimulation for 4,000 pulses followed by low-frequency right DLPFC stimulation for 1,000 pulses for a total stimulation time of approximately one hour per session. This protocol was chosen based on a recent meta-analysis (Brunoni et al., 2017) indicating that amongst the various treatment protocols, priming the low frequency right hemisphere stimulation with a high frequency left hemisphere stimulation led to the greatest efficacy for treatment of Major Depressive Episodes. Additionally, the overwhelming majority of the literature in TMS for depression targets the stimulation to DLPFC and the FDA has approved repetitive transcranial magnetic stimulation (rTMS) to DLPFC for the treatment of medication-resistant major depressive disorder (MDD).

The primary outcome will be change in depression severity from baseline to post-treatment. The primary analysis will be a comparison between the ICT-rTMS and sham groups. Secondary outcome measures utilized will include cognitive, quality of life, and emotional regulation measures, as well as imaging changes. Additional analyses will include durability of effects during the 6 months following treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-64
2. Current or former US military service member
3. Eligible for care at DoD facilities
4. Able to provide written, informed consent in English
5. History of concussive TBI:

   1. >6 months prior to consent
   2. Documented previously in medical records and/or as confirmed by the TBI Screener
6. Must meet Criterion A of the DSM-5 criteria for Major Depressive Disorder as determined by a trained assessor
7. Baseline MADRS >10

Exclusion Criteria:

1. Elevated risk of seizures:

   1. Prior history of unprovoked seizures other than within 24 hours of concussive TBI
   2. Family history of seizures
   3. History of TBI resulting in penetrating trauma based on the TBI Screener
   4. Presence of intracranial tumor or intraparenchymal hemorrhage based on the structural MRI scan
   5. Heavy alcohol consumption within 48 hours, prior to any treatment session
   6. Receiving tricyclic antidepressants or neuroleptics at doses that lower seizure threshold
2. Contraindications to awake 3T MRI without contrast:

   1. Ferromagnetic implants or metallic shrapnel
   2. Severe claustrophobia
   3. Unable to lie awake, supine, stationary, with reasonable comfort in the scanner for approximately 45 minutes
   4. Markedly distorted functional brain anatomy such that rsfMRI targeting cannot be performed
3. History of severe or recent uncontrolled heart disease
4. Presence of a cardiac pacemaker or intracardiac lines
5. Implanted neurostimulators and medication pumps
6. Presence of rapidly progressive illnesses such as late stage cancer, neurodegenerative conditions, major organ failure, etc.
7. History of Bipolar Disorder, Schizophrenia Spectrum Disorders, or Moderate/Severe Substance Use Disorders, with the exception of nicotine use disorders
8. Increased risk of suicide as clinically evaluated
9. Current evidence of substance-induced mood disorder, active psychosis, and/or depression secondary to general medical illness (other than TBI)
10. Concomitant or previous history of receiving open-label TMS, other neurostimulatory treatment, or electroconvulsive therapy
11. Pregnancy

    a. Female participants of childbearing potential must agree to use an effective method of birth control during the course of the study, or to remain abstinent from sex, to ensure they do not become pregnant during the course of the study
12. Unilateral or bilateral upper extremity amputation or other condition precluding motor threshold calibration
13. Any considerations that, in the opinion of the investigator, may adversely affect patient safety, participation, or the scientific validity of the data being collected (e.g., planned hospitalization halfway through the initial treatment period, limited life expectancy, etc.)

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2019-07-01 (Actual); Primary Completion 2020-10-27 (Actual); Study Completion 2020-10-27 (Actual)

PRIMARY OUTCOMES:
Improvement in Depressive Symptoms | Change between baseline, post-treatment (i.e., within 10 days of treatement completion), and 6-month follow-up
  Compare change in overall Montgomery-Asberg Depression Rating Scale (MADRS) scores between participants randomized to ICT-rTMS and those randomized to blinded sham stimulation. The overall score ranges from 0 to 60 with a higher overall score indicating more severe depression.

SECONDARY OUTCOMES:
Changes in Cognitive Function | Change between baseline, post-treatment (i.e., within 10 days of treatement completion), and 6-month follow-up
  Assess changes in cognitive function and emotion processing as measured by the Automated Neuropsychological Assessment Metric (ANAM).
Changes in TBI-related Symptoms | Change between baseline, post-treatment (i.e., within 10 days of treatement completion), and 6-month follow-up
  Assess changes in TBI-related symptoms as reflected by the TBI-QOL.
Changes in PTSD-related Symptoms | Change between baseline, post-treatment (i.e., within 10 days of treatement completion), and 6-month follow-up
  Assess changes in PTSD-related symptoms as reflected by the PTSD Checklist for DSM-5 (PCL-5).
Changes in Tinnitus-related Symptoms | Change between baseline, post-treatment (i.e., within 10 days of treatement completion), and 6-month follow-up
  To assess changes in tinnitus-related symptoms as reflected by the Mini Tinnitus Questionnaire (Mini TQ-12).
Frequency of Adverse Effects | Change between baseline, post-treatment (i.e., within 10 days of treatement completion), and 6-month follow-up
  Compare the frequency and severity of adverse effects between those randomized to ICT-rTMS and those randomized to blinded sham stimulation.
Changes in Psychotherapeutic Changes | Change between baseline, post-treatment (i.e., within 10 days of treatement completion), and 6-month follow-up
  Compare the number, dose, and/or type of adjunctive treatments undertaken by those randomized to ICT-rTMS as compared to those randomized to blinded sham stimulation.
Changes in Resting-state fMRI | Change between baseline, post-treatment (i.e., within 10 days of treatement completion), and 6-month follow-up
  Assess changes in resting-state functional connectivity using functional magnetic resonance imaging (fMRI).

CONTACTS AND LOCATIONS:
Overall Officials: David L Brody, MD, PhD, Principal Investigator — Center for Neuroscience and Regenerative Medicine (CNRM)
Locations (2):
- United States (2):
  - Walter Reed National Military Medical Center, Bethesda, Maryland
  - Fort Belvoir Community Hospital, Fort Belvoir, Virginia

IPD SHARING:
Plan to Share IPD: Yes
Coded data will be deposited into the following repositories: the Center for Neuroscience and Regenerative Medicine (CNRM) Data Repository and the Federal Interagency Traumatic Brain Injury Research (FITBIR) Database.
Time Frame: Following project completion, a summary of the results will be provided to the site.
Access Criteria: Access to the data located in the CNRM Repository and FITBIR database will be provided by the respective entities.

REFERENCES:
- [Background] Hacker CD, Laumann TO, Szrama NP, Baldassarre A, Snyder AZ, Leuthardt EC, Corbetta M. Resting state network estimation in individual subjects. Neuroimage. 2013 Nov 15;82:616-633. doi: 10.1016/j.neuroimage.2013.05.108. Epub 2013 Jun 2. PMID 23735260
- [Background] Brunoni AR, Chaimani A, Moffa AH, Razza LB, Gattaz WF, Daskalakis ZJ, Carvalho AF. Repetitive Transcranial Magnetic Stimulation for the Acute Treatment of Major Depressive Episodes: A Systematic Review With Network Meta-analysis. JAMA Psychiatry. 2017 Feb 1;74(2):143-152. doi: 10.1001/jamapsychiatry.2016.3644. PMID 28030740